CLINICAL TRIAL: NCT06789393
Title: Comparison of the Efficacy of Bupivacaine with and Without Dexmedetomidine As an Adjuvant on Penile Block for Postoperative Pain Relief in Pediatrics Undergoing Hypospadias Repair Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Almonaem Abd Alnazeer, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B+D hypospadias repair surgery
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hypospadias Repair Surgery
Keywords: penile block
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Penile block with bupivacaine 0.25% (0.2 ml/kg) plus dexmedetomidine (0.5 mcg/kg)
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine
- Group B (Placebo Comparator): Penile block with bupivacaine 0.25% (0.2 ml/kg) only
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive dexmedetomidine (0.5 mcg/kg).
  Arms: Group A
Drug: Bupivacaine — Penile block with bupivacaine 0.25% (0.2 ml/kg)

SUMMARY:
The main issue with pain management in children especially young children is the difficulty involved in evaluating it. When a patient's level of pain cannot be accurately assessed, effective analgesia cannot be prescribed. When children are not sufficiently treated for pain, stress hormones are released into their systems, resulting in increased catabolism, immunosuppression and hemodynamic instability .

Peripheral nerve blocks may be favored over neuroaxial blocks because they allow quicker mobilization after surgery.

Hypospadias results from abnormal development of the penis that leaves the urethral meatus proximal to its normal glanular position anywhere along the penile shaft, scrotum, or perineum. A spectrum of abnormalities, including ventral curvature of the penis (chordee), a hooded incomplete prepuce, and an abortive corpora spongiosum, are commonly associated with hypospadias. Surgical correction is typically performed during early childhood to restore normal appearance and function.

Penile block is a widely used regional anesthesia technique for hypospadias repair, It involves the administration of a local anesthetic around the penile nerve, providing effective pain relief during and after surgery. While effective, the duration of analgesia provided by a penile block with local anesthetics alone is often limited, necessitating the use of additional analgesics in the postoperative period.

Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with sedative, anxiolytic, and analgesic properties. It has been increasingly used as an adjuvant in regional anesthesia to prolong the duration of analgesia and reduce opioid consumption .

The addition of dexmedetomidine to local anesthetics has been shown to enhance the quality and duration of nerve blocks in various surgical settings but its efficacy in penile block for pediatric hypospadias repair has not been extensively studied.

the aim of the study To assess the duration of analgesia provided by the penile block with dexmedetomidine.

Timing and episodes of rescue analgesia consumption . To monitor and report any adverse effects associated with the use of dexmedetomidine such as hypotension and bradycardia

DETAILED DESCRIPTION:
The main issue with pain management in children especially young children is the difficulty involved in evaluating it. When a patient's level of pain cannot be accurately assessed, effective analgesia cannot be prescribed. When children are not sufficiently treated for pain, stress hormones are released into their systems, resulting in increased catabolism, immunosuppression and hemodynamic instability .

Peripheral nerve blocks may be favored over neuroaxial blocks because they allow quicker mobilization after surgery.

Hypospadias results from abnormal development of the penis that leaves the urethral meatus proximal to its normal glanular position anywhere along the penile shaft, scrotum, or perineum. A spectrum of abnormalities, including ventral curvature of the penis (chordee), a hooded incomplete prepuce, and an abortive corpora spongiosum, are commonly associated with hypospadias. Surgical correction is typically performed during early childhood to restore normal appearance and function.

Penile block is a widely used regional anesthesia technique for hypospadias repair, It involves the administration of a local anesthetic around the penile nerve, providing effective pain relief during and after surgery. While effective, the duration of analgesia provided by a penile block with local anesthetics alone is often limited, necessitating the use of additional analgesics in the postoperative period.

Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with sedative, anxiolytic, and analgesic properties. It has been increasingly used as an adjuvant in regional anesthesia to prolong the duration of analgesia and reduce opioid consumption .

The addition of dexmedetomidine to local anesthetics has been shown to enhance the quality and duration of nerve blocks in various surgical settings but its efficacy in penile block for pediatric hypospadias repair has not been extensively studied.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 7 years
* Scheduled for primary hypospadias repair under general anesthesia
* Parental consent obtained

Exclusion Criteria:

* - Known allergy to dexmedetomidine or other study medications .
* History of cardiovascular or respiratory disease.
* Active infection.
* History of developmental or mental retardation .
* Coagulation disorders.
* Parental refusal.

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
FLACC Pain score | 24 hours
  FLACC Pain score (Face,Leg,Activity,Cry,Consolability) in pediatric patients undergoing hypospadias repair(post-operative). A total score between 0 and 10 It will be measured at the recovery room and 2,6,12,24 hours posoprtatively

IPD SHARING:
Plan to Share IPD: Undecided